CLINICAL TRIAL: NCT00677365
Title: Phase II, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety, Tolerability and Efficacy of Three Dosage Regimens of MP-376 Solution for Inhalation Given for 28 Days to Stable CF Patients
Brief Title: Safety, Tolerability and Efficacy of MP-376 Given for 28 Days to Cystic Fibrosis (CF) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mpex-204; 2008-001728-30 (EudraCT Number)
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo inhaled either once or twice daily via the PARI eFlow nebulizer for 28 days
  Interventions: Drug: Placebo
- MP-376 120 mg QD (Experimental): MP-376 120 mg inhaled Once Daily (QD) via the PARI eFlow nebulizer for 28 days
  Interventions: Drug: MP-376
- MP-376 240 mg QD (Experimental): MP-376 240 mg inhaled QD bia the PARI eFlow nebulizer for 28 days
  Interventions: Drug: MP-376
- MP-376 240 mg BID (Experimental): MP-376 240 mg inhaled twice daily (BID) via the PARI eFlow nebulizer for 28 days
  Interventions: Drug: MP-376

INTERVENTIONS:
Drug: MP-376 — 3 dose regimens of MP-376 administered twice daily (BID) or once daily (QD) for 28 days
  Other Names: Levofloxacin Inhalation Solution; Aeroquin
  Arms: MP-376 120 mg QD; MP-376 240 mg BID; MP-376 240 mg QD
Drug: Placebo — same frequency as study drug using the same nebulizer
  Arms: Placebo

SUMMARY:
Patients with cystic fibrosis (CF) suffer from chronic infections of the lower respiratory tract that can be caused by one or multiple bacteria, including Pseudomonas aeruginosa, which has been particularly problematic to eradicate and been implicated as the major cause of morbidity and mortality in CF patients. Aerosol delivery of antibiotics directly to the lung increases the local concentrations of antibiotic at the site of infection resulting in improved antimicrobial effects compared to systemic administration. Bacterial resistance to current aerosol antibiotic treatments indicate a need for improved therapies to treat CF patients with pulmonary infections caused by multi-drug resistant Pseudomonas aeruginosa and other bacteria. High concentrations of MP-376 delivered directly to the lung are projected to have antimicrobial effects on even the most resistant organisms.

DETAILED DESCRIPTION:
This trial will be a double-blind, placebo-controlled study to evaluate the safety, tolerability and efficacy of levofloxacin administered as MP-376 of three dosage regimens given for 28 days by the aerosol route to CF patients.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria (selected):

* > 16 years of age
* Confirmed Diagnosis of Cystic Fibrosis
* Positive sputum culture for P. aeruginosa within the past 18 months
* Patients are able to elicit a forced expiratory volume in 1 second (FEV1) >/= 25% but </= 85% of predicted value at screening
* Have received at least 3 courses of inhaled antimicrobials over the preceding 12 months
* Clinically stable with no changes in health status within the last 30 days
* Able to reproducibly produce sputum and perform spirometry

Exclusion Criteria (selected):

* Use of any nebulized or systemic antibiotics within 30 days prior to baseline
* History of hypersensitivity to fluoroquinolones or intolerance with aerosol medication
* Evidence of acute upper within 10 days or lower respiratory infections within 30 days prior to dosing
* Creatine clearance < 50mg/ml, aspartate transaminase (AST), alanine transaminase (ALT) or total bilirubin >/= 3 x upper limit of normal (ULN) at Screening

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (50):
- United States (39):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Childrens Hospital, Los Angeles, California
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - Miami, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Oak Lawn, Illinois
  - Park Ridge, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Minneapolis, Minnesota
  - Las Vegas, Nevada
  - Morristown, New Jersey
  - Albany, New York
  - Valhalla, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Oklahoma CF Center, Oklahoma City, Oklahoma
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Memphis, Tennessee
  - San Antonio, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
- Germany (8):
  - Berlin
  - Essen
  - Frankfurt
  - Gerlingen
  - Gieben
  - Kiel
  - München
  - Tübingen
- Netherlands (3):
  - Amsterdam
  - Groesbeek
  - Rotterdam

REFERENCES:
- [Derived] Geller DE, Flume PA, Staab D, Fischer R, Loutit JS, Conrad DJ; Mpex 204 Study Group. Levofloxacin inhalation solution (MP-376) in patients with cystic fibrosis with Pseudomonas aeruginosa. Am J Respir Crit Care Med. 2011 Jun 1;183(11):1510-6. doi: 10.1164/rccm.201008-1293OC. Epub 2011 Feb 25. PMID 21471106

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo Group
- MP-376 120 mg QD: MP-376 120 mg Once Daily (QD) Group
- MP-376 240 mg QD: MP-376 240 mg Once Daily (QD) Group
- MP-376 240 mg BID: MP-376 240 mg Twice Daily (BID) Group
Period: Overall Study
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Started | 37 | 38 | 37 | 39
Completed | 35 | 37 | 35 | 36
Not Completed | 2 | 1 | 2 | 3
Not completed — Adverse Event | 2 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Other reason | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID | Total
Number analyzed (Participants) | 37 | 38 | 37 | 39 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (9.94) | 28.0 (6.86) | 27.5 (9.05) | 29.2 (9.98) | 28.7 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 16 | 14 | 66
  Male | 19 | 20 | 21 | 25 | 85
Region of Enrollment [Number; unit: Participants]
  United States | 30 | 32 | 30 | 32 | 124
  Europe | 7 | 6 | 7 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in P. Aeruginosa Density
Description: Patients were required to cough deeply and then spit sputum into a sterile container. The bacteria contained in the sputum sample was incubated in a laboratory and the number of P. aeruginosa colony forming units per gram of sputum (CFU/g) was determined. The difference in CFUs/g were then compared from baseline to the conclusion of the 28 day treatment period
Time Frame: from baseline to end of treatment (28 days)
Population: Modified Intent-to-Treat (MITT; patients who received at least one dose of study drug)
Measure: Least Squares Mean (Standard Error); unit: log10 CFU/g sputum
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Number analyzed (Participants) | 37 | 38 | 37 | 39
log10 CFU/g sputum | 0.23 (0.220) | -0.31 (0.227) | -0.31 (0.220) | -0.73 (0.222)
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; LS Mean Difference; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — Repeated Measure Model; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.54 to -0.38]

2. Secondary Outcome: Time to Administration of Other Anti-pseudomonal Antimicrobials
Description: Time to administration of other anti-pseudomonal antimicrobials in patients with at least one of the following: decreased exercise tolerance, increased cough, increased sputum/chest congestion, or decreased appetite; 25th percentile data reported
Time Frame: from baseline until final study visit (up to 56 days)
Population: MITT
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Number analyzed (Participants) | 37 | 38 | 37 | 39
days | 31 [29 to 43] | NA [32 to NA] — Not available; 25th percentile was not reached within the 56-day study duration | 56 [43 to NA] — Not available; The upper range of the confidence interval exceeds the 56-day study duration | 59 [57 to NA] — Not available; The upper range of the confidence interval exceeds the 56-day study duration
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; Hazard Ratio for need of anti-pseudomonal antimicrobials; Estimates are obtained from a Cox proportional hazards regression model including terms for treatment, region, baseline P.aeruginosa density (log10 ), highest baseline MIC of levofloxacin against P. aeruginosa (log2 ), and baseline percent predicted FEV1 (quartiles); Test type: Superiority or Other; p = 0.0007, Regression, Cox; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.09 to 0.52]

3. Secondary Outcome: Percent Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Percent change in the amount of air the patient could exhale in 1 second
Time Frame: from baseline to end of the 28-day treatment period (28 days)
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Number analyzed (Participants) | 37 | 38 | 37 | 39
Percent change | -2.36 (2.085) | 1.93 (2.114) | 2.56 (2.077) | 6.25 (2.081)
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; LS Mean Difference Between MP-376 240 mg and Placebo groups; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; Mean Difference (Final Values) = 8.61, 95% CI 2-sided [3.05 to 14.17]

4. Secondary Outcome: Change in FEV1 Percent Predicted
Description: Change in the predicted percent of air the patient could exhale in one second
Time Frame: from baseline to the end of the treatment 28-day treatment period (28 days)
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Number analyzed (Participants) | 37 | 38 | 37 | 39
Percent | -2.39 (2.370) | 1.96 (2.402) | 3.10 (2.361) | 8.55 (2.358)
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; LS Mean Difference Between Placebo and MP-376 240 mg BID groups; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = 10.94, 95% CI 2-sided [4.63 to 17.25]

5. Secondary Outcome: Changes in Respiratory Domain Scores of Cystic Fibrosis Questionnaire - Revised (CFQ-R)
Description: Change in the score from 0 to 100 that a patient reports for their respiratory symptoms in the CFQ-R. An increase in score illustrates an improvement in symptoms. An increase of 4 or more is considered clinically significant
Time Frame: from baseline to the end of the 28-day treatment period (28 days)
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Number analyzed (Participants) | 37 | 38 | 37 | 39
units on a scale | -0.44 (2.715) | 2.00 (2.728) | 0.31 (2.689) | 4.06 (2.690)
Statistical Analysis 1: Comparison: Placebo vs MP-376 240 mg BID; LS Mean Difference from MP-376 240 mg BID to placebo groups; Test type: Superiority or Other; p = 0.2174, Mixed Models Analysis; Mean Difference (Final Values) = 4.50, 95% CI 2-sided [-2.68 to 11.67]

6. Secondary Outcome: Changes in Susceptability Patterns of Isolated Organisms
Description: All isolates of P. aeruginosa cultures grown from patient sputum samples were evaluated to see whether the minimum concentration of levofloxacin needed to inhibit growth of the bacteria (i.e., minimum inhibitory concentration; MIC) had increased; 2. The MIC50 and MIC90 values were calculated as the 50th percentile value and the 90th percentile value, respectively. Note that percentile values between dilution values were rounded up to the nearest dilution value
Time Frame: from baseline until the end of the 28-day treatment period (28 days)
Population: MITT
Measure: Number; unit: ug/mL
Units Other Than Participants: Isolates
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Number analyzed (Participants) | 37 | 38 | 37 | 39
Number analyzed (Isolates) | 140 | 152 | 148 | 152
ug/mL
  Baseline Minimum Inhibitory Concentration (MIC)50 | 4 | 4 | 4 | 4
  Day 28 MIC for 50% (MIC50) | 4 | 4 | 4 | 4
  Baseline MIC for 90% (MIC90) | 16 | 32 | 16 | 16
  Day 28 MIC90 | 8 | 16 | 16 | 32

ADVERSE EVENTS:
Arm/Group | Placebo | MP-376 120 mg QD | MP-376 240 mg QD | MP-376 240 mg BID
Serious Adverse Events (participants affected / at risk) | 4/37 | 1/38 | 4/37 | 4/39
Other Adverse Events (participants affected / at risk) | 28/37 | 33/38 | 32/37 | 33/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | MP-376 120 mg QD (N=38) | MP-376 240 mg QD (N=37) | MP-376 240 mg BID (N=39)
Disease progression (General disorders) | 3 (3) | 0 (0) | 4 (4) | 3 (3) — Pulmonary exacerbation
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | MP-376 120 mg QD (N=38) | MP-376 240 mg QD (N=37) | MP-376 240 mg BID (N=39)
Dysgeusia (Nervous system disorders) | 1 (1) | 14 (15) | 18 (19) | 13 (14) — Taste complaint
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 9 (9) | 10 (12) | 10 (11)
Disease progression (General disorders) | 10 (12) | 4 (4) | 8 (9) | 7 (7) — Pulmonary exacerbation
Headache (Nervous system disorders) | 0 (0) | 7 (8) | 2 (2) | 4 (4)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 3 (3) | 5 (6) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 2 (2) | 6 (6)
Pharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Chest Discomfort (General disorders) | 3 (3) | 0 (0) | 2 (2) | 4 (5)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No